CLINICAL TRIAL: NCT06865027
Title: Effect of Arterial Carbon Dioxide Levels on Cerebral Blood Flow and Cerebral Autoregulation in Steep Trendelenburg Position During Robot-assisted Prostatectomy, and Its Effect on Postoperative Cognition - A Clinical Blinded Randomized Trial
Brief Title: The Effect of Arterial Carbon Dioxide Levels on Cerebral Blood Flow and Cerebral Autoregulation in the Steep Trendelenburg Position During Robot-assisted Prostatectomy, and Its Effect on Postoperative Cognition
Acronym: TILTDOWN-3
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Signe Søvik, Professor, Senior Consultant, PhD, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REK:744921; 2022088 (Other Grant/Funding Number: South-Eastern Norway Regional Health Authority)
Record Dates: First submitted 2025-02-26; First posted 2025-03-07 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Intracranial Pressure; Circulation System; Cerebral Perfusion Pressure; Cognitive Function
Keywords: RALP surgery; Postoperative cognitive disorder; Cerebral perfusion pressure; Cerebral circulation; Cerebral autoregulation; Trendelenburg position; Robot-assisted laparoscopic prostatectomy; Transcranial Doppler ultrasound
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Intervention Model Description: Clinical double blinded randomized interventional study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant and investigator are blinded. The anesthesia providers are not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypercapnia (Other): PaCO2: 6.4-7.0 kPa
  Interventions: Other: Ventilation strategy
- Normocapnia (Other): PaCO2: 5.0-5.5 kPa
  Interventions: Other: Ventilation strategy

INTERVENTIONS:
Other: Ventilation strategy — The selected PaCO2 targets are:
  Normocapnia: PaCO2: 5.0-5.5 kPa Hypercapnia: PaCO2: 6.4-7.0 kPa
  The adjustments on the ventilator needed to achieve these targets will be administered by the anesthetic nurse and attending anesthesiologist and held within the following limitations:
  Tidal volume: 4 - 8ml ml/kg IBW Inspiratory pressure 5-30 cm H2O Respiration rate 10-18 per minute PEEP 5-10 mmHg
  *IBW: 50 + 0.91 (height in centimeters - 152.4) Peep, I:E ratio, and FiO2 will be administered at the anesthetic nurse's and the anesthesiologist's discretion.
  Other Names: normocapnia; hypercapnia

SUMMARY:
Patients scheduled for robot-assisted prostatectomy will be randomized to either high or low concentrations of carbon dioxide in the blood. This will be managed by applying different ventilation strategies during anesthesia.The levels will be distinctly different.

The investigators will assess whether different concentrations of carbon dioxide in blood results in different brain blood flow levels and different intracranial pressure during laparascopic surgery in the head-down tilted position. The investigators also will assess if different carbon dioxide level will manifest in different cognitive abilities in the two study groups, measured on day 1 post-surgery.

DETAILED DESCRIPTION:
Detailed Description: The carotid artery carries blood into the brain. Therefore, blood flow levels in the carotid artery may be used to assess brain perfusion. Brain perfusion is carefully regulated by the body, to ensure that the brain always receives enough oxygen and nutrients. During prostate surgery using laparoscopic techniques, the patient lies tilted on the operating table, with their head markedly lower than their legs. The investigators aim to study the effect on cerebral blood flow of a head-down tilted body position in combination with anesthesia and laparoscopic surgery, and particularly how cerebral blood flow is influenced by the participants' breathing pattern. The study aims to achieve insights that may be used to improve the treatment of vulnerable surgical patients, such as those with cerebrovascular disease or severe heart disease.

Anesthesia and surgery will proceed as usual, with the exception that the respiratory support the participants receive during the surgery will be adjusted as described below. The participants will receive standard monitoring of heart rate, blood pressure, and blood oxygen levels. Before surgery, the anesthesia team will per routine insert two plastic cannulas into the left arm for administering medication, and a plastic cannula into the participant's left wrist for close monitoring of the participant's blood pressure.

Study participants will undergo four additional steps:

1. Before surgery, an anesthesiologist will insert a thin plastic cannula into a superficial vein on the side of the neck. The cannula is the same type as the ones used on the arm and has a diameter of 1.1 mm. The purpose of this cannula is to measure the pressure of the blood returning from the brain to the heart. The procedure involves brief, moderate pain associated with the needle insertion. The plastic cannula will be removed before the participant wakes up from anesthesia.
2. Just before and during surgery, a trained anesthesiologist will perform ultrasound measurements on the right side of the participant's neck, temple, and the outside of the eyelid. Each measurement lasts 4-5 minutes. This will not prolong the time spent in the operating room. The measurements will cause no discomfort.
3. All patients undergoing prostate removal with robotic surgery receive respiratory support with a ventilator during anesthesia. In this study, the investigators will adjust the ventilator to control the carbon dioxide (CO2) levels towards either the lower or upper normal range for CO2. A blinded randomization will determine the group assignment. Regardless of which group a participant is assigned to, their CO2 level will be maintained within a range routinely used during anesthesia and considered completely safe.

In the project, the investigators will collect and record participant information. The investigators will store recordings of the participants' pulse, blood pressure, breathing depth and rhythm, levels of oxygen and CO2 in the participants' blood, medication doses used during surgery, and results of blood tests taken during surgery. From the participants' medical records, the investigators will retrieve and record the participants' age, gender, height, weight, whether the participants have chronic diseases, and which regular medications the participants use.

Cognitive tests of reaction time and problem-solving abilities will be administered a few days before and one day after surgery.

Receiving information about an illness, undergoing a surgical procedure, receiving general anesthesia, peroperative CO2 levels, body position during robotic surgery, and postoperative pain medication all affect the body physically and may trigger stress and anxiety. The investigators want to assess this impact using a well-established method that tests reaction time through five exercises on an iPad. The method has been developed for use in patients. Those participating in the study will be asked to perform this test at the outpatient clinic a few days before surgery and one day after surgery.

ELIGIBILITY:
Inclusion Criteria: Males 55-80 years old, accepted by surgeon and attending anesthesiologist for RALP surgery.

Exclusion Criteria:

* Poorly controlled hypertension (resting BP >165/90 on pre-study consult).
* Emphysema of the lung.
* Previous spontaneous pneumothorax.
* Cerebrovascular disease. Including but not limited to previous SAH, EDH, SDH, hemorrhage from AVM, known AVM and stenosis in carotid or cerebral arteries.
* Intracranial malignancy or metastases from primary cancer.
* Significant cardiovascular disease (NYHA class III or IV).
* Renal failure grade 4 or 5 (estimated GFR <30).
* Anatomical hinders for performing ultrasound of the right carotid artery or middle cerebral artery.
* Primary language other than Scandinavian.
* Diagnosed dementia of any subtype.

Ages: 55 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
ICA flow | day of surgery
  Changes in cerebral blood flow (ml/s) during surgery

SECONDARY OUTCOMES:
Cognitive performance | 5 days pre-surgery and 1 day post-surgery
  Measurements of cognitive performance by CANTAB tests (Cambridge Cognition, England)
Cerebral perfusion pressure | Day of surgery
  Estimated ICP (mmHg) minus Mean arterial pressure (mmHg).
Cardiac index (L/min) | Day of surgery
  Measured by LidCO arterial pulse contour analysis

CONTACTS AND LOCATIONS:
Overall Officials: Signe Søvik, Professor, MD, PhD, Study Director — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lørenskog, Norway

IPD SHARING:
Plan to Share IPD: No
Any sharing of patient-level data from this study would have to be pre-approved by the Regional Committee for Medical and Health Research Ethics in South-Eastern Norway as well as by the Personal Data Protection Officer at Akershus University Hospital